CLINICAL TRIAL: NCT06026878
Title: Gemcitabine Combined With Nimotuzumab and Toripalimab as Induction Treatment Followed by Chemoradiotherapy for Locally Advanced Nasopharyngeal carcinoma-a Multicenter, Randomized Controlled Study
Brief Title: GNT Induction Treatment in Locally Advanced NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, clinical professor of department of radiation oncology of XiJing hospital, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFMMUChina
Record Dates: First submitted 2023-08-29; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; nimotuzumab; toripalimab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- gemcitabine, nimotuzumab and toripalimab induction treatment (Experimental): Gemcitabine at a dose of 1 g per square meter of body-surface area on days 1 and 8 every 3 weeks for two cycles.
  nimotuzumanb 400mg every 3 weeks for two cycles. toripalimab 240mg every 3 weeks for two cycles.
  Interventions: Drug: gemcitabine,nimotuzumab, toripalimab
- gemcitabine and cisplatin (Active Comparator): Gemcitabine at a dose of 1 g per square meter of body-surface area on days 1 and 8 and cisplatin at a dose of 80 mg per square meter on day 1 were administered intravenously once every 3 weeks for two cycles.
  Interventions: Drug: gemcitabine, cisplatin

INTERVENTIONS:
Drug: gemcitabine,nimotuzumab, toripalimab — same as before
  Other Names: GNT
  Arms: gemcitabine, nimotuzumab and toripalimab induction treatment
Drug: gemcitabine, cisplatin — same as before
  Other Names: GP
  Arms: gemcitabine and cisplatin

SUMMARY:
The goal of this clinical trial is to compare overall response rate between gemcitabine, nimotuzumab and toripalimab as induction treatment and gemcitabine combined with cisplatine in paitents with locally advanced nasopharyngeal carcinoma. It aims to answer whether gemcitabine, nimotuzumab and toripalimab as induction treatment show non-inferiority compared to GP induction chemotherapy. Participants will be randomly divided into two induction treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old.
2. Pathologically or cytologically confirmed stage III-IVB nasopharyngeal keratinizing squamous cell carcinoma or non-keratinizing squamous cell carcinoma.
3. Patients suitable for radical radiochemotherapy.
4. ECOG PS score of 0-1.
5. According to the RECIST 1.1 criteria, there is at least one measurable lesion. Basic hematological parameters are normal: white blood cell count ≥4×10^9/L; absolute neutrophil count ≥1.5×10^9/L; platelets ≥100×10^9/L; hemoglobin ≥90 g/L.
6. Basically normal renal function: serum creatinine ≤1.5×ULN or creatinine clearance rate (CrCl) > 60 mL/min (using the Cockcroft-Gault formula): For females: CrCl = (140-age) x weight (kg) x 0.85 / (72 x Scr mg/dl) For males: CrCl = (140-age) x weight (kg) x 1.00 / (72 x Scr mg/dl)
7. Basically normal liver function: serum total bilirubin ≤1.5×ULN; aspartate aminotransferase (AST) ≤2.5×ULN; alanine aminotransferase (ALT) ≤2.5×ULN.
8. Signed written informed consent.

Exclusion Criteria:

1. Patients who have previously undergone immunotherapy or targeted therapy.
2. Participated in any other interventional clinical trials within 30 days before screening.
3. History of other malignancies (except for cured skin basal cell carcinoma).
4. History of primary immunodeficiency.
5. Presence of uncontrolled concurrent diseases (such as heart failure, severe lung disease, severe liver disease, mental disease, etc.).
6. Known HIV infection, active viral hepatitis, or tuberculosis.
7. Major surgery within 90 days before the first dose of the study drug, or planned surgery.
8. Allergic to the drugs used in this protocol or their components.
9. Pregnant (confirmed by blood or urine HCG tests) or breastfeeding women, or those of childbearing age unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last trial treatment.
10. The investigator believes the subject is not suitable for this study.
11. Unwilling to participate in this study or unable to sign the informed consent form.
12. Live vaccinations within 30 days of dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | three weeks after induction therapy
  the proportion of patients who achieve complete response and partial response after induction therapy

SECONDARY OUTCOMES:
2-year overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  2-year survival rate of patients enrolled in this study
2-year distant metastasis-free survival | From date of randomization until the date of distant metastasis or last follow-up time,, whichever came first, assessed up to 100 months
  2-year distant metastasis-free survival rate of patients enrolled in this study
2-year local regional recurrence-free survival | From date of randomization until the date of local and/or lymph node recurrence or last follow-up time,, whichever came first, assessed up to 100 months
  2-year local regional recurrence-free survival rate of patients enrolled in this study

OTHER OUTCOMES:
adverse events | through study completion, an average of 1 year
  treatment-related adverse events during treatment and follow-up time

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No